CLINICAL TRIAL: NCT03307265
Title: Impact of the Use of a Weighted Jacket on the Balance (While Walking or Standing) of Patients With a Balance Disorder.
Brief Title: Impact of the Use of a Weighted Jacket on the Balance of Patients With a Balance Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernard Dachy (Other)
Responsible Party: Sponsor-Investigator, Bernard Dachy, Head of neurology department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUB-Weighted jacket
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Balance; Distorted
Keywords: Weighted Jacket; Balance disorder; Equilibrium disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imbalance correction (Experimental)
  Interventions: Device: Personalized weighted jacket
- Control (Active Comparator)
  Interventions: Device: Control jacket

INTERVENTIONS:
Device: Personalized weighted jacket — Patients in this group will wear a jacket with weights (1,5 to 2% of the total body mass) strategically placed in order to correct their imbalance.
  Arms: Imbalance correction
Device: Control jacket — Patients in this group will wear a jacket with weights (200 grams maximum) evenly distributed.
  Arms: Control

SUMMARY:
The aim of the study is to test whether wearing a weighted jacket can help improve the balance distortion of patients with neurologic pathologies.

The center of mass of the patient will be analyzed in order to determine the direction in which the imbalance is most important. Weights will be placed accordingly in a jacket in order to correct the imbalance. In the experimental group, weights will represent 1.5 to 2% of the patient body mass. In the control group, the investigators will use weights of 200 grams maximum, placed evenly on both sides of the jacket. Patients will wear the jacket for 2 consecutive hours.

After wearing the jacket for 2 hours, data similar to those recorded at the beginning of the experiment will be taken again, namely the determination of the center of mass and of the deviations caused by the imbalance.

A final series of tests will take place approximately one week after wearing the jacket, to determine if there are any residual effects.

ELIGIBILITY:
Inclusion Criteria:

* good level of French understanding
* be able to walk a minimum distance of 10 meters with or without rod/walker
* walk 10 meters in more than 12 seconds.
* have a diagnosis of Multiple Sclerosis, Parkinson's, or any other neurological pathology that could cause balance disorders
* be able to endure at least 2 hours of tests, interviews or medical care.
* score of more than 8 seconds at the time up and go (TUG), less than 24 points out of 28 in the Tinetti test

Exclusion Criteria:

* the patient underwent a period of exacerbation of his pathology in the last two months (especially for multiple sclerosis patients)
* chronic back pain
* poor eyesight (not be able to perform the tests)
* osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Imbalance | Data measured after 2 hours of jacket utilisation
  The side towards which the patient is more likely to be unbalanced is determined by an interactive balance linked to the Wii-fit.
Time Up and Go | Data measured after 2 hours of jacket utilisation
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Tinetti test | Data measured after 2 hours of jacket utilisation
  The Tinetti test or score is a simple, reproducible way of assessing the risk of falls.
Berg balance scale | Data measured after 2 hours of jacket utilisation
  The Berg balance scale includes 14 tests that assess static balance and dynamic balance.

SECONDARY OUTCOMES:
Imbalance | 1 week after jacket utilisation
  The side towards which the patient is more likely to be unbalanced is determined by an interactive balance linked to the Wii-fit.
Time Up and Go | 1 week after jacket utilisation
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Tinetti test | 1 week after jacket utilisation
  The Tinetti test or score is a simple, reproducible way of assessing the risk of falls.
Berg balance scale | 1 week after jacket utilisation
  The Berg balance scale includes 14 tests that assess static balance and dynamic balance.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No